CLINICAL TRIAL: NCT03526471
Title: Prospective, Single-arm Study to Assess the Safety and Performance of the Omega™ Left Atrial Appendage (LAA) Occluder in Patients With Non-Valvular Atrial Fibrillation and High Bleeding Risk
Brief Title: Omega™ Left Atrial Appendage (LAA) Occluder in Patients With Non-Valvular Atrial Fibrillation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vascular Innovations Co. Ltd. (Industry)
Collaborators: MedPass International (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LAAC
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2020-08-27 (Actual); Status verified 2020-08

CONDITIONS: Atrial Fibrillation
Keywords: Left Atrial Appendage; Non-valvular atrial fibrillation; High Bleeding Risk
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Left Atrial Appendage (LAA) Occluder (Experimental): Left Atrial Appendage (LAA) Occluder
  Interventions: Device: Omega™ Left Atrial Appendage (LAA) Occluder

INTERVENTIONS:
Device: Omega™ Left Atrial Appendage (LAA) Occluder — catheter delivery of Omega device in the left atrial appendage

SUMMARY:
Atrial fibrillation is associated with increased risk of stroke mostly because of clot formation in the left atrial appendage, a small alcove in the left atrium heart chamber. Plugging this appendage with an implantable plug type device, which is placed via a catheter painlessly in the femoral vein, has been proven to be a reliable alternative to the standard anti-clotting medication in a number of recent international trials. The Omega device is a new design of such a plug, made from biocompatible and compressible nitinol and fabric.

Up to 195 patients will be enrolled in Europe, assuming that enrolment will stop once the Omega™ device has been successfully implanted in 150 evaluable patients.

The primary performance endpoint of the study is LAA closure (defined as complete seal or efficient seal with a peri-device leak ≤ 5 mm) at 60 days (+/- 15 days) visit documented by transoesophageal echocardiogram (TEE/TOE) with colour flow Doppler.

DETAILED DESCRIPTION:
This is a single arm study to assess the safety and performance of the Omega™ Left Atrial Appendage (LAA) Occluder in patients with Non-valvular atrial fibrillation (NVAF) and high bleeding risk.

The study will be conducted in accordance with the ISO standard ISO 14155 (Clinical investigation of medical devices for human subjects - Good clinical practice) and other legal requirements as applicable.

The primary performance endpoint of the study is LAA closure (defined as complete seal or efficient seal with a peri-device leak ≤ 5 mm) at 60 days (+/- 15 days) visit documented by transoesophageal echocardiogram (TEE/TOE) with colour flow Doppler.

The primary safety endpoint of the study is device-related complications (serious adverse events [SAEs]) through 60 days (+/- 15 days) post-procedural.

Following consent a number of assessments will be undertaken prior to the procedure to ensure the study eligibility criteria are met. These assessments include; medical history, physical exams, ECG, blood tests, transthoracic echocardiogram, transesophageal echocardiogram and cardiac CT.

The implant procedure will usually be performed under general anaesthetic. A thin catheter is inserted in the femoral vein in the right groin area and advanced under X-Ray guidance to the right atrium, then a very small needle is used to cross through to the left atrium to allow the delivery catheter to place the Omega in the Appendage, guided by both X-Ray and transesophageal echo. A medication regimen for endocarditis prophylaxis anticoagulation is recommended post procedure.

Following discharge, patients will be seen again at 60 days, 6 months and 12 months to collect data for the primary performance endpoint (by TTE or TEE) and safety endpoints (mRS, stroke/TIA assessments, and ECG).

An interim analysis is planned following the collection of 60 day data for the first 10 patients implanted with the device. An additional interim analysis will be performed following the collection of 60 days (+/- 15 days) data for the first 50 patients implanted with the device.

Final analysis will be performed once all 150 subjects have been implanted with the device and completed the study to further document and confirm the safety and effectiveness of the device.

ELIGIBILITY:
Inclusion Criteria:

1. 60 years of age or older
2. Documented paroxysmal, persistent, or permanent non-valvular atrial fibrillation (AF)
3. At increased risk of stroke or systemic embolism defined as CHADS2 score > 2 or a CHA2DS2-VASc score > 3
4. Deemed, by investigator, to be unsuitable or contraindicated for long term oral anticoagulation therapy due to high bleeding risk
5. To have suitable anatomy for percutaneous LAA occlusion procedure with a single Omega™ device based on CT scan evaluation
6. Able and willing to comply with the required medication regimen post-device implant
7. Able to understand and willing to provide written informed consent to participate in the study
8. Able to and willing to return for required follow-up visits and examinations.

Exclusion criteria:

1. Requires long-term oral anticoagulation therapy for any indication other than atrial fibrillation
2. Contraindicated for or allergic to aspirin, clopidogrel, warfarin or novel oral anticoagulant (NOAC) use
3. Has undergone surgical atrial septal defect (ASD) repair or has an ASD closure device implanted
4. Has undergone surgical patent foramen ovale (PFO) repair or has a PFO closure device implanted
5. Implanted with a mechanical heart valve prosthesis thus requiring long term oral anticoagulation
6. Has any contraindications for a percutaneous catheterization procedure (e.g. subject is too small to accommodate the transoesophageal echocardiogram (TEE/TOE) probe or required catheters, or subject has active infection or bleeding disorder)
7. Stroke or transient ischemic attack (TIA) within 90 days prior to implant procedure
8. Underwent any cardiac or non-cardiac intervention or surgery within 30 days prior to implant, or intervention or surgery is planned within 60 days after implant procedure
9. Myocardial infarction (MI) within 90 days prior to implant
10. New York Heart Association Class IV Congestive Heart Failure
11. Left ventricular ejection Fraction (LVEF) <30%
12. Symptomatic carotid artery disease (defined as >50% reduced diameter with symptoms of ipsilateral transient or visual TIA evidenced by amaurosis fugax, ipsilateral hemispheric TIAs or ipsilateral stroke); if subject has a history of carotid stent or endarterectomy the subject is eligible if there is >50% reduced diameter
13. Reversible cause of AF (i.e. secondary thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures)
14. History of idiopathic or recurrent venous thromboembolism requiring long term oral anticoagulation
15. Left atrial appendage is obliterated or surgically ligated
16. Resting heart rate >110 bpm
17. Thrombocytopenia (defined as < 70,000 platelets/mm3) or anaemia with haemoglobin concentration of < 10 g/dl (i.e. anaemia as determined by the investigator which would require transfusion)
18. Actively enrolled or plans to enrol in a concurrent clinical study in which the active treatment arm may confound the results of this trial
19. Active endocarditis or other infection producing bacteraemia
20. Subject has a known malignancy or other illness where life expectancy is less than 2 years
21. Impaired renal function with eGFR <40 ml/min/1.73 m2
22. More than mild hepatic failure, i.e. ALT, AST, or Alkalic Phosphatase >2× upper limit of normal

Echocardiographic Exclusion Criteria:

1. Intracardiac thrombus - including LAA - visualized by echocardiographic imaging
2. Existing circumferential pericardial effusion >2mm
3. Significant mitral valve stenosis (i.e. mitral valve area <1.5 cm2)
4. High risk patent foramen ovale (PFO), defined as an atrial septal aneurysm (atrial septal excursion >15mm; excursion defined as maximal protrusion of the ASA beyond the plane of the atrial septum during cardiac cycle) or large shunt (substantial passage of bubbles, i.e. >25, within 3 cardiac cycles from appearing in the right atrium)
5. Complex atheroma with mobile plaque of the descending aorta and/or aortic arch
6. Cardiac tumour
7. LAA anatomy cannot accommodate an Omega™ device (as per IFU)
8. Placement of the device would interfere with any intracardiac or intravascular structure.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
LAA closure | at 60 days (+/- 15 days)
  Complete seal or efficient seal with a peri-device leak ≤ 5 mm documented by transoesophageal echocardiogram (TEE/TOE) with colour flow Doppler.
Device-related complications | through 60 days post-procedure
  Serious adverse event criteria set out in the protocol and being assessed as related to the study device.

SECONDARY OUTCOMES:
Procedure-related complications | 1 to 6 days post-procedure
  Meeting the serious adverse event criteria set out in the protocol and being assessed as related to the study procedure.
Major bleeding | From procedure to 12 months
  Defined as ≥ BARC 3 bleed
Ischemic stroke | From procedure to 12 months
  Confirmed by Neurologic assessment and appropriate CT/MR imaging
Systemic embolism | From procedure to 12 months
  Confirmed by appropriate imaging.
Pericardial effusion/tamponade | From procedure to 12 months
  Per protocol
Technical success | At implant
  Composite of: Occlusion of the LAA, No device-related complications, No leak >5mm on colour Doppler Transesophageal Echocardiography (TEE),
Procedural success | At procedure
  Composite of: Technical success, No procedure-related complications except uncomplicated (minor) device embolization resolved by percutaneous retrieval during the procedure without surgical intervention or damage to surrounding cardiovascular structures.

CONTACTS AND LOCATIONS:
Overall Officials: Aidan Mulloy, Study Director — Eclipse Medical Ltd.
Locations (2):
- Rigshospitalet, Copenhagen, Denmark
- Chulalongkorn University, Pathum Wan, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No